CLINICAL TRIAL: NCT04474262
Title: Efficacy of Albumin Plus Midodrine v/s Albumin Alone in Reducing Incidence of Paracentesis Induced Circulatory Dysfunctions in ACLF Patients-A Randomized Controlled Trial.
Brief Title: Efficacy of Albumin Plus Midodrine v/s Albumin Alone in Reducing Incidence of Paracentesis Induced Circulatory Dysfunctions in ACLF Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-ACLF-06
Record Dates: First submitted 2020-07-01; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Albumins; Midodrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin with placebo (Active Comparator): Group A will be given albumin 8g/l of ascitic tap along with placebo for 7 days. Standard albumin therapy will continue (40gm/week)
  Interventions: Biological: Albumin; Other: Placebo
- Albumin with Midodrine (Experimental): GROUP B will be given midodrine 7.5 mg to 10 mg tds (keeping the target MAP above 70 mmhg)for 7 days plus albumin same as in other group.
  Interventions: Biological: Albumin; Drug: Midodrine Oral Tablet

INTERVENTIONS:
Biological: Albumin — Albumin will be 8g/l of ascitic tap. Standard albumin therapy will continue (40gm/week)
Drug: Midodrine Oral Tablet — Midodrine 7.5 mg to 10 mg TDS (keeping the target MAP above 70 mmHg).
  Arms: Albumin with Midodrine
Other: Placebo — Placebo
  Arms: Albumin with placebo

SUMMARY:
The patients with ACLF having Ascites who require ascitic tapping will undergone ascitic tapeither under albumin cover alone or with midodrine. The patient will be monitored for complication and changes of PICD. Study analysis will be done with primary objective being reduction in incidence of PICD.

DETAILED DESCRIPTION:
OBJECTIVE:

Primary objective: Incidence of Paracentesis induced circulatory dysfunction in patients undergoing modest volume paracentesis (MVP) (>3 and <5 litres) with midodrine plus 25% albumin v/s 25% albumin infusion alone at day 7

Secondary objective:

* Change in systolic, diastolic and mean BP at day 3 and 6
* Increase in plasma renin activity at day 6
* Incidence of Hyponatremia, HE and AKI at day 3 and 6
* Predictors of Paracentesis induced circulatory dysfunction
* Predictors of 28 day survival.

Methodology :

Patients with Acute on chronic liver failure having grade III ascites will be given either albumin or albumin plus midodrine. Midodrine will be started 4 hrs before tap to achieve target MAP. Ascitic tapping will be followed by vital monitoring and monitoring of vital parameters along with measurement of changes in s. rennin at day 3 and 6.

* All patient will be undergo complete physical examination and complete clinical history will be recorded.
* Baseline cbc,LFT,KFT and INR level will be sent on day 1 along with baseline s. renin levels
* Those eligible will be randomised in to two groups
* GROUP A will be given albumin 8g/l of ascitic tap during tap along with placebo for 7 days.
* GROUP B will be given midodrine 7.5 mg to 12.5 mg tds (keeping the target MAP above 70 mmhg)for 7 days plus albumin same as in other group.

Study Population: Patients of acute on chronic liver failure who are admitted to and attending the OPD at ILBS.

Study Design: Randomized controlled trial Study Period:NOV 2019 to march 2019

Sample Size:

Considering incidence of PICD in albumin group is 30% and reduction to 10% by adding midodrine with alpha =5%, and power of study being 80%. No. of cases in each group- 66 Total-132 Furthur with 10% dropout we need to enroll 150 cases (75 in each group) randomly allocated in two groups by block randomization method with block size of 5.

* Intervention: This RCT will be conducted at ILBS New Delhi between Dec 2019 and March 2021
* Monitoring and assessment:
* All patient will be undergo complete physical examination and complete clinical history will be recorded.
* Baseline cbc,LFT,KFT and INR level will be sent on day 1 along with baseline s. renin levels
* Those eligible will be randomised in to two groups
* GROUP A will be given albumin 8g/l of ascitic tap along with placebo for 7 days. Standard albumin therapy will continue (40gm/week)
* GROUP B will be given midodrine 7.5 mg to 10 mg tds (keeping the target MAP above 70 mmhg)for 7 days plus albumin same as in other group.

Expected outcome of the project:

Primary:

* Incidence of PICD at day 3 and day6

Secondary:

* Changes in hemodynamic parameters at 1, 3 and 6 hour, Day 3, Day 6 post paracentesis
* Increase in plasma renin activity at Day 3, Day 6
* Incidence of Hyponatremia, HE and AKI at day 3 and 6

ELIGIBILITY:
Inclusion Criteria:

- ACLF patients (as per APASL definition) with grade II/III ascites

Exclusion Criteria:

1. Age < 18 or >75 years
2. Hepatocellular carcinoma
3. Extrahepatic portal vein obstruction
4. Non cirrhotic ascites
5. Serum creatinine >1.5mg/dl
6. Refractory septic shock
7. Beta blockersPortal vein thrombosis
8. Grade 3-4 HE
9. Pregnancy or Lactation
10. Active variceal bleed
11. Respiratory, cardiac, renal failure
12. Uncontrolled hypertension
13. Severe coagulopathy
14. Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of PICD (Paracentesis Induced Circulatory Dysfunction) | Day 3
Incidence of PICD (Paracentesis Induced Circulatory Dysfunction) | Day 6

SECONDARY OUTCOMES:
Changes in Mean Arterial Pressure (MAP) post paracentesis. | 1 hour
Changes in Heart Rate post paracentesis. | 1 hour
Changes in Mean Arterial Pressure (MAP) post paracentesis. | 3 hours
Changes in Heart Rate post paracentesis. | 3 hours
Changes in Mean Arterial Pressure (MAP) post paracentesis. | 6 hours
Changes in Heart Rate post paracentesis. | 6 hours
Changes in Mean Arterial Pressure (MAP) post paracentesis. | Day 3
Changes in Heart Rate post paracentesis. | Day 3
Changes in Mean Arterial Pressure (MAP) post paracentesis. | Day 6
Changes in Heart Rate post paracentesis. | Day 6
Change in plasma renin activity in both groups | Day 3
Change in plasma renin activity in both groups | Day 6
Incidence of Hyponatremia in both groups | Day 3
Incidence of Hyponatremia in both groups | Day 6
Incidence of Hepatic Encephalopathy in both groups | Day 3
Incidence of Hepatic Encephalopathy in both groups | Day 6
Incidence of Acute Kidney Injury in both groups | Day 3
Incidence of Acute Kidney Injury in both groups | Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided